CLINICAL TRIAL: NCT01602471
Title: An Exploratory, Phase II, Open Label, Single-Center, Non-Randomized Study Of [F-18] RGD-K5 Positron Emission Tomography (PET) In Participants With Carotid Artery Stenosis
Brief Title: [F-18] RGD-K5 Positron Emission Tomography (PET) in Participants With Carotid Artery Stenosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to develop the product in collaboration
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: K5-C200
Record Dates: First submitted 2011-09-14; First posted 2012-05-21 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-07

CONDITIONS: Carotid Stenosis
Keywords: Endarterectomy; K5-C200; RGD-K5; angiogenesis; Carotid CT Angiogram
MeSH Terms: conditions — Carotid Stenosis | interventions — 18F-RGD-K5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F-18]RDG-K5 (Experimental): [F-18]RDG-K5 was administred and PET scan performed
  Interventions: Drug: [F-18]RDG-K5

INTERVENTIONS:
Drug: [F-18]RDG-K5 — Approximately fifteen (15) patients with carotid artery stenosis > 69% will undergo an endarterectomy and will be imaged under PET/CT with [F-18]RGD-K5
  Other Names: RGD-K5; K5; [F-18]RGD-K5 PET scan; RGD-K5 PET scan; K5 PET scan

SUMMARY:
This trial will be the first trial for the Investigation Product (IP), [F-18]RGD-K5 for carotid plaque imaging and will be conducted as a Phase II trial since this compound has already been tested in humans for phase I and phase II imaging. All study results will be evaluated and analyzed in order to consider the design for future clinical trials.

DETAILED DESCRIPTION:
This investigation will be conducted as a Phase II, open-label, single-center, non-randomized study. The study is planned to be conducted at one Investigative site in the United States. The information collected under this exploratory, Phase II study will not be used for diagnostic purposes, to assess the participant's response to therapy, or for clinical management of the participant. This will be a pilot prospective cohort study where the increased expression of integrin may be seen on the F-18 RGD-K5 PET imaging scans looking at carotid plaque in participants with carotid artery stenosis.

Each completed study participant will undergo one to three visits, including one eligibility study visit, the Computed Tomography (CT) angiogram of the carotid visit (if necessary), the [F-18] RGD-K5 PET imaging visit, and a 24 hour follow up phone call or visit.

Procedures: Informed consent (ICF), eligibility blood labs, collection of demographic information and medical history, physical examination, vital signs, 12-lead Electrocardiograms (ECGs), dosing with [F-18]RGD-K5, PET imaging scan, 24 hour follow up to collect adverse events, and plaque immunohistochemical characterization after Carotid Endarterectomy (CEA).

ELIGIBILITY:
Inclusion Criteria:

* Participant is a female or male of any race / ethnicity >18 years old at the time of the investigational product administration
* Participant or participant's legally acceptable representative provides written informed consent
* Participant is capable of complying with study procedures
* Participant has known carotid artery stenosis of >69% luminal diameter as based on carotid ultrasound and who is deemed to be a surgical candidate for endarterectomy as determined by the vascular surgeon
* Participant has had a carotid ultrasound and the report is available for collection
* Participant has had or is scheduled to have a carotid CT angiogram for plaque localization within 30 days of signing ICF (or else scheduled Carotid CT angiogram) CTA must be performed on a separate day and prior to the investigational PET procedure)
* Participant has consented to have an endarterectomy
* Participant will be scheduled for an investigational [F-18]RGD-K5 PET/CT scan within 4 weeks prior to endarterectomy
* Participant must have renal function values as defined by laboratory results within the following ranges:
* Serum creatinine ≤ 1.5 mg/dL
* Estimated glomerular filtration rate (eGFR) ≥ 45mL/min

Exclusion Criteria:

* Participant is nursing
* Participant is pregnant
* Participant has been involved in an investigative, radioactive research procedure within the past 14 days
* Participant has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality
* Participant has a history or current evidence of any condition, therapy, lab abnormality that, in the opinion of the study investigator or treating physicians might confound the results of the study or poses an additional risk to the participants by their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balaji Tamarappoo, MD, PhD, Principal Investigator — The Cleveland Clinic; Edward Aten, MD, Study Director — President, Certus International
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants enrolled, four complete and one withdrawal prior to receiving the investigational product. Study was terminated early by the sponsor.
Period: Overall Study
Arm/Group | [F-18]RDG-K5
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Five participants enrolled, four complete and one withdrawal prior to receiving the investigational prodcut. Study was terminated early by the sponsor.
Arm/Group | [F-18]RDG-K5
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 70.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: [F-18]RDG-K5 Uptake by Carotid Plaque on PET Scan
Description: Based on the small sample size and lack of IHC analyses, no efficacy conclusions can be drawn from this study.
Time Frame: Participants will be followed for an average of 6 weeks
Arm/Group | [F-18]RDG-K5
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | [F-18]RDG-K5
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No